CLINICAL TRIAL: NCT04799015
Title: A Randomized Study of Dexamethasone as Adjuvant Therapy for Acute Post-traumatic Headache
Brief Title: Dexamethasone for Post Traumatic Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-12625
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Dexamethasone; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 10mg IV + metoclopramide 10mg IV
  Interventions: Drug: Dexamethasone; Drug: Metoclopramide 10mg
- Placebo (Placebo Comparator): Placebo IV + metoclopramide 10mg IV
  Interventions: Drug: Metoclopramide 10mg

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10mg IV
  Arms: Dexamethasone
Drug: Metoclopramide 10mg — Metoclopramide 10mg IV

SUMMARY:
This is a randomized study of intravenous metoclopramide + intravenous dexamethasone versus intravenous metoclopramide for patients with acute post-traumatic headache.

ELIGIBILITY:
Inclusion Criteria:

Meet International Classification of Headache Disorders criteria for acute post-traumatic headache as follows:

* Traumatic injury to the head has occurred
* Headache has developed within 7 days of injury to the head
* Headache is not better accounted for by another diagnosis (e.g., migraine or tension-type headache)
* The headache must be rated as moderate or severe in intensity at the time of initial evaluation

Exclusion Criteria:

* More than ten days have elapsed since the head trauma
* Headache has already been treated with an anti-dopaminergic medication
* Medication allergies
* Contra-indications including pheochromocytoma, seizure disorder, Parkinson's disease, use of MAO inhibitors, and use of anti-rejection transplant medications

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Frequency Moderate or Severe headache after Emergency Department (ED) discharge | Up to 48 hours after ED discharge
  Headache intensity will be rated based on the International Headache Society (IHS) 4-point scale. Using this scale participants will verbalize whether their headache intensity is "severe," "moderate," "mild," or "none." The percentage of patients reporting a headache intensity level of either "moderate" or 'severe" will be summarized by study arm. Between-group difference along with 95% confidence intervals will be reported. Patients who use an analgesic or abortive headache medication during the 48 hour period will be considered an outcome failure and their results will not be included in the analysis.

SECONDARY OUTCOMES:
Sustained headache relief | 48 hours after ED discharge
  Sustained headache relief will be defined as the number of patients achieving a headache intensity of "mild" or "none" and who maintain that level for 48 hours after ED discharge without the use of rescue medication. The percentage of patients reporting both headache intensity level of either "moderate" or 'severe" will be summarized by study arm.
Post concussive symptoms | 48 hours after ED discharge
  Post concussive symptoms at 48 hours will be assessed using the Sport Concussion Assessment Tool (SCAT) Post Concussion Symptom Scale (PCSS). Using the validated SCAT PCSS patients rate the severity of 22 concussive symptoms on a 7-point Likert scale ranging from 0 ("none") to 6 ("severe") yielding an overall possible scoring range of 0-132. Higher SCAT PCSS scores are indicative of more severe level of post-concussive symptoms. Results will be summarized by study arm using basic descriptive statistics.
Post concussive symptoms | 7 days after ED discharge
  Post concussive symptoms at 7 days will be assessed using the Sport Concussion Assessment Tool (SCAT) Post Concussion Symptom Scale (PCSS). Using the validated SCAT PCSS patients rate the severity of 22 concussive symptoms on a 7-point Likert scale ranging from 0 ("none") to 6 ("severe") yielding an overall possible scoring range of 0-132. Higher SCAT PCSS scores are indicative of more severe level of post-concussive symptoms. Results will be summarized by study arm using basic descriptive statistics.
Use of Rescue medication | Duration of ED admission, up to 3-4 days
  Use of rescue medication will be defined as the number of patients administered any analgesic medication or headache abortive medication while in the ED. The number of patients using rescue medication will be summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No